CLINICAL TRIAL: NCT01009723
Title: Early Prediction Of Preterm Delivery By Measurement Of Maternal Serum Markers
Brief Title: Preterm Delivery Risk Prediction by Measurement of Prenatal Serum Screening Markers
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Esoterix Genetic Laboratories, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: GGPS0001
Record Dates: First submitted 2009-11-05; First posted 2009-11-09 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Preterm Delivery
Keywords: Preterm delivery; preterm labor; maternal-fetal care; maternal serum screening biomarkers; alphafetoprotein; AFP; human chorionic gonadotropin; hCG; unconjugated estriol; Inhibin A; pregnancy associated plasma protein; PAPP-A; maternal screening
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples from the study subjects
Oversight: Data Monitoring Committee: No

SUMMARY:
This protocol seeks to longitudinally collect blood samples from a cohort of pregnant women. The biological specimens will be used to determine the predictive power of biochemical markers routinely used in Down syndrome screening in the assessment of patient's risk of preterm delivery.

DETAILED DESCRIPTION:
The study will investigate whether the levels of individual maternal serum screening biomarkers, their combinations or temporal changes in the level can be associated with an increased risk of preterm delivery. Blood samples at three time points in pregnancy will be collected from the study participants. The first two blood draws will be timed to coincide with the first and second trimester maternal serum testing. The third blood draw will coincide with the screening for gestational diabetes. Pregnancy outcome information will be collected from the physicians and linked to the subject samples.

Subject samples from a case-control patient group will be analyzed by the serum screening biochemical assay. Statistical analyses will be performed to achieve the study objectives.

NOTE: This study is recruiting in Florida, USA. The laboratory data coordination is being performed in Massachusetts, USA and New Mexico, USA. New study locations will be identified on an ongoing basis.

ELIGIBILITY:
Inclusion Criteria:

* The participant understands the nature of the study and its requirements. To this end, we will require that the participants have command of the English language.
* The participant consents to and signs the approved consent form.
* The participant is 18 years of age or older.
* The participant has a singleton pregnancy.
* The participant is planning on continuing the pregnancy.
* The participant has intent to clinically test for Down syndrome risk.
* The participant consents to the study at the first trimester of her pregnancy.
* The participant understands the nature of the study and its requirements. To this end, we will require that the participants have command of either the English or Spanish language.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population of the US
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Esoterix Genetic Laboratories, LLC
Locations (2):
- United States (2):
  - Integrated Genetics, Westborough, Massachusetts
  - Integrated Genetics, Santa Fe, New Mexico

REFERENCES:
- [Background] Chitayat D, Farrell SA, Huang T, Meier C, Wyatt PR, Summers AM. Double-positive maternal serum screening results for down syndrome and open neural tube defects: An indicator for fetal structural or chromosomal abnormalities and adverse obstetric outcomes. Am J Obstet Gynecol. 2002 Sep;187(3):758-63. doi: 10.1067/mob.2002.125240. PMID 12237660
- [Background] Lepage N, Chitayat D, Kingdom J, Huang T. Association between second-trimester isolated high maternal serum maternal serum human chorionic gonadotropin levels and obstetric complications in singleton and twin pregnancies. Am J Obstet Gynecol. 2003 May;188(5):1354-9. doi: 10.1067/mob.2003.278. PMID 12748511